CLINICAL TRIAL: NCT03396133
Title: Assessment of Portable Remote Health Monitor Using the Snap to Symptomatic Arrhythmia
Brief Title: Efficacy of Snap on Symptomatic Arrhythmia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, principal investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 009
Record Dates: First submitted 2017-12-07; First posted 2018-01-10 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Arrhythmia
Keywords: Snap; symptomatic arrhythmia; diagnosis; follow-up
MeSH Terms: conditions — Arrhythmias, Cardiac; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snap group (Experimental): individuals in this arm used Snap according to the instruction on time and screened at the symptomatic
  Interventions: Diagnostic Test: Snap
- RC group (No Intervention): patients in the RC arm accepted normal methods

INTERVENTIONS:
Diagnostic Test: Snap — screen, transmission, and analysis ECG automated
  Arms: Snap group

SUMMARY:
Participants in the Snap arm were instructed to undertake once-day recording and transmission of a 30-second single-lead iECG trace to a secure server, plus additional submissions if symptomatic over a 3-month period. Snap traces were analyzed by an automated analysis software and cardiologists. Clinical review and appropriate care was arranged for those clinically significant arrhythmia. Patients in the RC group were followed up as normal methods including ECG, Holter.

DETAILED DESCRIPTION:
Individuals with symptomatic arrhythmia without known arrhythmia were recruited.

Participants were required to have access to the internet via WiFi and to be able to operate the Snap system after simple instruction. Written consent was obtained, and eligible participants were randomized (1:1) to an intervention (Snap) group or RC group.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic arrhythmia

Exclusion Criteria:

* can not use the Snap instrument and Sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the ability of handheld device with remote interpretation to screen for arrhythmia | 3-month
  Participants in Snap group acquired ECG once od according to the rules and transmitted ECG immediately once symptom appeared between 3-month. Patients in the routine treatment (RT) group were administrated normal diagnostic techniques. At 3-month, compared the incidence atrial arrhythmia(atrial premature beats and atrial tachycardia) and ventricula arrhythmia(ventricular premature beats and ventricular tachycardia) between two groups.

SECONDARY OUTCOMES:
Evaluating the patients' quality of life | 3-month
  Using RAND 36-Item Short Form Health Survey (SF-36) 1.0 Questionnaire items assessed the quality of life of participants. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are: vitality, physical functioning, bodily pain, general, health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. The total scale ranges from 35 to 145. The higher the total score, the better the patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Jian Li, PHD, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Jin-Shuang Li, MD, Principal Investigator — Suqian People's Hospital of Nanjing Drum Tower Hospital Group; Liang-Hong Ying, MD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - Dyno, Nanjing, Jiangsu
  - the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Halcox JPJ, Wareham K, Cardew A, Gilmore M, Barry JP, Phillips C, Gravenor MB. Assessment of Remote Heart Rhythm Sampling Using the AliveCor Heart Monitor to Screen for Atrial Fibrillation: The REHEARSE-AF Study. Circulation. 2017 Nov 7;136(19):1784-1794. doi: 10.1161/CIRCULATIONAHA.117.030583. Epub 2017 Aug 28. PMID 28851729